CLINICAL TRIAL: NCT02203695
Title: Phase II Randomized Placebo-Controlled Double-Blind Study of Salvage Radiation Therapy (SRT) Plus Placebo Versus SRT Plus Enzalutamide in Men With High-Risk PSA-Recurrent Prostate Cancer After Radical Prostatectomy
Brief Title: Randomized Salvage Radiation Therapy Plus Enzalutamide Post Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Astellas Pharma Inc (Industry); Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: J1454; IRB00030471 (Other: JHMIRB)
Record Dates: First submitted 2014-06-16; First posted 2014-07-30 (Estimated); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: Salvage Radiation Therapy (SRT); Enzalutamide
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SRT plus Enzalutamide (Experimental): Arm 2 (experimental): (SRT) Salvage radiation therapy (Three dimensional conformal radiation therapy (3D-CRT)/IMRT [Intensity-modulated radiation therapy]) 66.6-70.2 Gy as 1.8 Gy M-F for 37-39 fx PLUS Enzalutamide (MDV3100) 160 mg PO once daily for 6 months (2 months prior to SRT, 2 months during SRT and 2 months following SRT)
  Interventions: Drug: Enzalutamide
- SRT plus placebo (Placebo Comparator): Arm 1 (control): Salvage radiation therapy (3D-CRT (Three dimensional conformal radiation therapy)/IMRT (Intensity-modulated radiation therapy)) 66.6-70.2 Gy given 1.8 Gy M-F for 37 -39 fx PLUS Placebo PO daily for 6 months (2 months prior to SRT, 2 months during SRT and 2 months following SRT)
  Interventions: Radiation: SRT

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide (MDV3100) 160 mg PO once daily for 6 months (2 months prior to SRT, 2 months during SRT and 2 months following SRT)
  Other Names: XTANDI
  Arms: SRT plus Enzalutamide
Radiation: SRT — Salvage radiation therapy (3D-CRT (Three dimensional conformal radiation therapy)/IMRT) 66.6-70.2 Gy given 1.8 Gy M-F for 37 -39 fx
  Other Names: Salvage Radiation Therapy
  Arms: SRT plus placebo

SUMMARY:
The primary hypothesis of this study is that outcomes for patients with biochemically recurrent prostate cancer following radical prostatectomy will be improved by the addition of enzalutamide for 6-months compared to standard-of-care salvage radiation therapy to allow for further study in the definitive phase III setting. This study builds on the prior success of high-dose bicalutamide (for 24 months) when combined with salvage external radiation therapy (XRT), while using a newer more potent anti-androgen for a shorter duration of time (6 months) in an effort to minimize adverse effects.

DETAILED DESCRIPTION:
Enzalutamide is a second-generation androgen receptor signaling inhibitor that significantly prolongs survival in patients with metastatic castration-resistant prostate cancer who have received prior docetaxel chemotherapy 35,36. Enzalutamide has demonstrated activity in cells that overexpress the androgen receptor. Unlike previous androgen receptor blocker (ARB) agents, Enzalutamide does not display any agonist properties and blocks translocation of the ligand-receptor complex into the nucleus preventing DNA binding 33. Enzalutamide is an oral agent that is generally well tolerated and does not require concurrent steroid administration, which makes it an ideal candidate for combination with salvage radiation therapy (SRT).

Finally, provocative preliminary Phase II data presented at the American Society of Clinical Oncology (ASCO) 2013 by M. Smith and colleagues assessed the efficacy and safety of 25-weeks (~6-mos) of enzalutamide alone in prostate cancer of all stages who had never received hormone therapy; presenting with non-castrate testosterone levels ( 230 ng/dL). Enzalutamide alone for 6-mos achieved a high PSA response rate with efficacy similar to castration, but .in contrast to castration, bone mineral density (BMD) remained stable and metabolic variables were not substantially impacted.

The trial described here differs from Radiation Therapy Oncology Group (RTOG) 96-01, RTOG 05-34 and RADICALS in several ways. First, the eligibility criteria are stricter; less favorable patients have been selected. Second, short-term ARB is being tested, while in RTOG 96-01 and RADICALS long-term ARB of 2-years was examined. Finally, and most importantly, we are testing the second generation ARB agent, enzalutamide, alone in combination with SRT as opposed to RTOG 05-34 and RADICALS which use androgen deprivation (AD).

This trial is not intended to address the efficacy of SRT alone over observation. The complete response rate (a drop in PSA to undetectable levels) after SRT is 70%-80% and durable responses are observed in 30%-40% of patients. For these reasons, it is not feasible or appropriate to randomize men between observation and SRT. The more important issue is whether the proportion of durable responses is increased by altering the therapeutic approach, such as the use of enhanced ARB using enzalutamide.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and Health Insurance Portability and Accountability Act (HIPPA) authorization for the release of personal health information.
* Males aged 18 years of age and above
* Patients must have adenocarcinoma of the prostate gland
* Patients must have received primary treatment with radical prostatectomy.
* Patients must have evidence of biochemical (PSA) relapse after prostatectomy
* Patients must have PSA within study range
* Patients must have non-metastatic (M0) disease, as defined by a lack of metastases seen on CT scan of the chest/abdomen/pelvis and whole-body radionuclide 99Technetium (Tc) bone scan, (or sodium fluoride PET scan) taken within 3 months of study entry.
* Patients must have had node negative (pN0) disease found at the time of surgery.
* Patients must have non-castrate levels of serum testosterone levels within study range.
* Patients must not have previously received hormonal therapy (LHRH agonist, antiandrogen, or both), with the exception of neoadjuvant or adjuvant hormones given in conjunction with prostatectomy.
* Patients must have Eastern Cooperative Oncology Group (ECOG)performance status of 0-1, and life expectancy greater 3 years.
* Patients must have laboratory test results within the certain ranges
* Patients must be disease-free from prior malignancies for greater than 3 years, with the exception of non-melanoma skin cancers and superficial urothelial cancers.
* Patients must have the ability to swallow the study drug whole as a tablet or capsule.
* Throughout study, male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration or per local guidelines where these require additional description of contraceptive methods.
* Throughout the study, patients must use a condom if having sex with a pregnant woman.

Exclusion Criteria:

* Currently active second malignancy
* Primary treatment with radiation therapy.
* Radiographic or clinical evidence of local-regional tumor recurrence,
* Concurrent use of other antiandrogens, estrogen-like agents, or 5a-reductase inhibitors.
* Use of systemic corticosteroids equivalent to prednisone (inhaled corticosteroids are permitted).
* Concurrent use of other anti-cancer agents or treatments.
* Serious concurrent medical illnesses (including uncontrolled major cardiac, pulmonary, Child-Pugh C liver or psychiatric diseases) or active major infections (including HIV, Hepatitis A-C).
* Clinically significant cardiovascular disease including:

  * Myocardial infarction within 6 months of Screening visit.
  * Uncontrolled angina within 3 months of Screening visit.
  * Congestive heart failure (within certain ranges)
  * History of clinically significant ventricular arrhythmias
  * Prolonged corrected QT interval
  * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place.
  * Hypotension within certain ranges
  * Uncontrolled hypertension within certain ranges
* Medications which lowers seizure threshold.
* History of seizure or any condition that may predispose to seizure including, but not limited to underlying brain injury, stroke, primary brain tumors, brain metastases, or alcoholism. Also, history of loss of consciousness or transient ischemic attack within 12months of enrollment (Day 1 visit).
* Patients taking medications that may have adverse interactions with enzalutamide

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-03-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Song, M.D., Principal Investigator — The SKCCC at Johns Hopkins
Locations (9):
- United States (9):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Lafayette, Indiana
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Oregon Health Sciences University, Portland, Oregon
  - University of Utah - Huntsman Cancer Center, Salt Lake City, Utah

REFERENCES:
- [Derived] Tran PT, Lowe K, Tsai HL, Song DY, Hung AY, Hearn JWD, Miller S, Proudfoot JA, Deek MP, Phillips R, Lotan T, Paller CJ, Marshall CH, Markowski M, Dipasquale S, Denmeade S, Carducci M, Eisenberger M, DeWeese TL, Orton M, Deville C, Davicioni E, Liauw SL, Heath EI, Greco S, Desai NB, Spratt DE, Feng F, Wang H, Beer TM, Antonarakis ES. Phase II Randomized Study of Salvage Radiation Therapy Plus Enzalutamide or Placebo for High-Risk Prostate-Specific Antigen Recurrent Prostate Cancer After Radical Prostatectomy: The SALV-ENZA Trial. J Clin Oncol. 2023 Feb 20;41(6):1307-1317. doi: 10.1200/JCO.22.01662. Epub 2022 Nov 11. PMID 36367998
- [Derived] Kapoor R, Deek MP, McIntyre R, Raman N, Kummerlowe M, Chen I, Gaver M, Wang H, Denmeade S, Lotan T, Paller C, Markowski M, Carducci M, Eisenberger M, Beer TM, Song DY, DeWeese TL, Hearn JW, Greco S, DeVille C, Desai NB, Heath EI, Liauw S, Spratt DE, Hung AY, Antonarakis ES, Tran PT. A phase II randomized placebo-controlled double-blind study of salvage radiation therapy plus placebo versus SRT plus enzalutamide with high-risk PSA-recurrent prostate cancer after radical prostatectomy (SALV-ENZA). BMC Cancer. 2019 Jun 13;19(1):572. doi: 10.1186/s12885-019-5805-z. PMID 31196032

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SRT Plus Enzalutamide | SRT Plus Placebo
Started | 43 | 43
Completed | 41 | 42
Not Completed | 2 | 1
Not completed — Patient withdrew consent | 1 | 1
Not completed — Started non-study treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SRT Plus Enzalutamide | SRT Plus Placebo | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Full Range); unit: Years] | 69 [51 to 82] | 66 [52 to 81] | 67 [51 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 43 | 43 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 37 | 40 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 43 | 86

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Freedom of PSA (Prostate Specific Antigen) Progression
Description: The primary efficacy endpoint is the rate of Freedom-from-PSA-progression (FFPP) at 2-years. FFPP is defined as the time from randomization to the date of PSA progression. A subject who does not have PSA progression at the time of the analysis will be censored at the last date of PSA measurement.
Time Frame: From time of randomization to date of PSA progression, approximately 2 years.
Measure: Number; unit: Percent of patients with no progession
Arm/Group | SRT Plus Enzalutamide | SRT Plus Placebo
Number analyzed (Participants) | 43 | 43
Percent of patients with no progession | 84 | 66

2. Secondary Outcome: Number of Participants With Local Recurrence
Description: Local recurrence within the radiation field (confirmed pathologically) at 2-years
Time Frame: 2 years from end of radiation therapy
Measure: Number; unit: Participants with local recurrence
Arm/Group | SRT Plus Enzalutamide | SRT Plus Placebo
Number analyzed (Participants) | 43 | 43
Participants with local recurrence | 0 | 0

3. Secondary Outcome: Metastatic Free Survival Rate
Description: Metastasis-free survival (MFS) rates at 2 years. Metastasis-free survival will be defined as the time from the date of registration to date of evidence of systemic disease on bone scan or cross sectional imaging or death, which occurs first. Number of participants with a metastasis event at 2 years is reported.
Time Frame: 2 years from the time of registration
Measure: Number; unit: participants
Arm/Group | SRT Plus Enzalutamide | SRT Plus Placebo
Number analyzed (Participants) | 43 | 43
participants | 0 | 1

4. Secondary Outcome: How Well Participants Tolerate Treatment Assessed by European Organization for Research & Treatment of Cancer Quality of Life (Questionnaire (EORTC-QLQ-P25)
Description: The European Organization for the Research and Treatment of Cancer (EORTC-QLQ-P25) quality of life questionnaire, Prostate Cancer Module. Uses a 4-point Likert scale, with responses ranging from "not at all" to "very much" for sexual symptoms and treatment related symptoms. Domain scores range 0 to 100, with higher scores reflecting either more symptoms (urinary, bowel, hormonal treatment-related symptoms) or higher levels of activity or functioning (sexual).
Time Frame: Baseline, End of Treatment (180 Days) and 6 Months Post-treatment
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SRT Plus Enzalutamide | SRT Plus Placebo
Number analyzed (Participants) | 11 | 11
score on a scale
  Baseline-Sexual Symptoms | 53.70 (44.56) | 41.67 (10.39)
  End of Treatment (180 days) -Sexual Symptoms: number analyzed (Participants) | 10 | 9
  End of Treatment (180 days) -Sexual Symptoms | 59.72 (38.32) | 42.22 (11.52)
  6 Months Post-treatment-Sexual Symptoms: number analyzed (Participants) | 7 | 4
  6 Months Post-treatment-Sexual Symptoms | 35.19 (22.45) | 35.19 (3.21)
  Baseline-Treatment related Symptoms | 9.09 (24.85) | 4.04 (3.59)
  End of treatment (180 days) -Treatment related Symptoms: number analyzed (Participants) | 10 | 9
  End of treatment (180 days) -Treatment related Symptoms | 14.44 (8.77) | 3.09 (2.92)
  6 Months Post-treatment-Treatment Related Symptoms: number analyzed (Participants) | 7 | 4
  6 Months Post-treatment-Treatment Related Symptoms | 11.11 (6.42) | 1.39 (2.78)

5. Secondary Outcome: How Well Participants Tolerate Treatment Assessed by the Functional Assessment of Cancer Therapy-Prostate (FACT-P).
Description: The Functional Assessment of Cancer Therapy (FACT-P), assesses the health-related quality of life in men with prostate cancer. The score is the sum of all 5 domain scores and ranges from 0 to156 where higher scores represent better quality of life.
Time Frame: Baseline, End of Treatment (180 Days) and 6 Months Post-treatment
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SRT Plus Enzalutamide | SRT Plus Placebo
Number analyzed (Participants) | 11 | 11
score on a scale
  Baseline | 126.15 (13.06) | 129 (15.54)
  End of Treament (180 Days): number analyzed (Participants) | 10 | 9
  End of Treament (180 Days) | 123.40 (12.02) | 124.33 (21.90)
  6 months Post-Treament: number analyzed (Participants) | 7 | 4
  6 months Post-Treament | 126.86 (13.69) | 137.25 (4.03)

6. Secondary Outcome: How Well Participants Tolerate Treatment Assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30).
Description: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire score range is from 0 to 100. A higher score indicates a better level of functioning or quality of life.
Time Frame: Baseline, End of Treatment (180 Days) and 6 Months Post-treatment
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SRT Plus Enzalutamide | SRT Plus Placebo
Number analyzed (Participants) | 11 | 11
score on a scale
  Baseline-Physical Functioning | 92.22 (10.68) | 100. (0.00)
  End of Treatment - (180 Days) Physical Functioning: number analyzed (Participants) | 10 | 9
  End of Treatment - (180 Days) Physical Functioning | 95.33 (8.92) | 97.04 (6.76)
  6 Months Post-treatment - Physical Functioning: number analyzed (Participants) | 7 | 4
  6 Months Post-treatment - Physical Functioning | 92.22 (10.68) | 100. (0.00)

7. Secondary Outcome: How Well Participants Tolerate Treatment Assessed by Sexual Health Inventory in Men (SHIM) Questionnaire.
Description: Quality of life (QoL) tool used to determine participant tolerability of treatment assessed by Sexual Health inventory in Men (SHIM). The questionnaire includes 5-items, and provides a total score from 1 to 25, with higher scores indicating better erectile function and lower scores indicating more severe erectile dysfunction.
Time Frame: Baseline, End of Treatment (180 Days) and 6 Months Post-treatment
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SRT Plus Enzalutamide | SRT Plus Placebo
Number analyzed (Participants) | 11 | 11
score on a scale
  Baseline | 7.36 (9.16) | 12.27 (10.97)
  End of Treatment (180 days): number analyzed (Participants) | 10 | 9
  End of Treatment (180 days) | 4.8 (7.55) | 10.89 (9.48)
  6 months Post-Treatment: number analyzed (Participants) | 7 | 4
  6 months Post-Treatment | 6.14 (9.46) | 16.25 (10.5)

8. Secondary Outcome: Feasibility of Achieving Stated Accrual
Description: Anticipated accrual of participants versus actual reported enrollment. The goal is 48 in each arm.
Time Frame: 2 years
Population: The Overall Number of Participants analyzed represents the goal of 48 participants in each arm.
Measure: Count of Participants; unit: Participants
Arm/Group | SRT Plus Enzalutamide | SRT Plus Placebo
Number analyzed (Participants) | 48 | 48
Participants | 43 | 43

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | SRT Plus Enzalutamide | SRT Plus Placebo
All-Cause Mortality (participants affected / at risk) | 2/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 43/43 | 43/43
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SRT Plus Enzalutamide (N=43) | SRT Plus Placebo (N=43)
nocturia (Nervous system disorders) | 13 (13) | 13 (13)
lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
erectile dysfunction (Nervous system disorders) | 8 (8) | 9 (9)
hypertension (General disorders) | 9 (9) | 5 (5)
fall (General disorders) | 0 (0) | 1 (1)
humerus fracture (General disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 28 (28) | 23 (23)
urinary frequency/urgency (Renal and urinary disorders) | 17 (17) | 21 (21)
diarrhea (Gastrointestinal disorders) | 13 (13) | 11 (11)
breast and nipple pain (General disorders) | 11 (11) | 0 (0)
sexuality alteration (General disorders) | 12 (12) | 9 (9)
urinary incontinence (Renal and urinary disorders) | 4 (4) | 10 (10)
Anorexia (Psychiatric disorders) | 5 (5) | 1 (1)
hemmorrhoids (Gastrointestinal disorders) | 9 (9) | 5 (5)
hot flashes (Endocrine disorders) | 7 (7) | 6 (6)
hyperglycemia (Endocrine disorders) | 5 (5) | 4 (4)
nausea (Gastrointestinal disorders) | 6 (6) | 2 (2)
pain (due to XRT) (General disorders) | 6 (6) | 4 (4)
Proctitis (General disorders) | 6 (6) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT02203695/Prot_SAP_000.pdf